CLINICAL TRIAL: NCT02156726
Title: Observational Study of Low Dose FCR in the Treatment of Elderly/Comorbid Patients With Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma: The Q-lite Project
Brief Title: Observational Study of Low Dose FCR in Elderly/Comorbid CLL/SLL: The Q-lite Project
Acronym: Q-lite
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Czech CLL Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: Q-lite
Record Dates: First submitted 2014-05-24; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; fludarabine; rituximab; elderly; comorbid; FCR; CIRS
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Receptors, Fc; fludarabine; Cyclophosphamide; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low dose FCR in Elderly/Comorbid CLL: low dose FCR
  Interventions: Drug: low-dose FCR

INTERVENTIONS:
Drug: low-dose FCR — FCR with attenuated dose of fludarabine and cyclophosphamide
  Other Names: Fludarabine; Cyclophosphamide; Rituximab

SUMMARY:
FCR (fludarabine, cyclophosphamide, rituximab) combination is currently accepted as the gold standard in treatment of younger and physically fit CLL patients. These excellent results, however, cannot be generally applied to the whole CLL population. This is because the median age at diagnosis of CLL lies between 65 and 72 years and patients older than 65 years in fact account up to 50%-75 % of the CLL population. Nevertheless, such population is considerably underrepresented in most of the large clinical trials in CLL/SLL. Therefore, it is not clear whether elderly/comorbid patients could profit from newer treatment approaches such as purine analog combinations or chemoimmunotherapy. Several publications demonstrated unacceptable toxicity of full-dose FC/FCR in elderly CLL patients. However, regimens using attenuated doses of fludarabine and cyclophosphamide showed promising efficacy and low toxicity.

DETAILED DESCRIPTION:
The objective of this observational study is to provide additional data to confirm the safety profile and efficacy of low dose FCR for CLL patients treated in clinical practice.

Specific data of interest are: comorbid concitions, concomitant medication, CLL characteristics, prior treatment regimens, adverse events, reasons for discontinuation low dose FCR, overal response rates, complete response rate, progression-free survival, overall survival.

This is an observational, non-interventional, medical record review study in CLL patients. A total of 200 patients with CLL who have been previously treated with low dose FCR will be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of CLL or SLL
* previously treated by low dose FCR for active disease requiring treatment per IWCLL criteria
* dose reduction of fludarabine and cyclophosphamide due to age, comorbid conditions, or reduce creatinine clearance

Exclusion Criteria:

* patients treated with low dose FCR within prospective clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CLL or SLL deemed unfit for full-dose FCR. Both untreated and relapsed/refractory setting.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-10 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 8 months
  Toxicity assessed by CTCAE criteria (myelotoxicity, infections, etc.)

SECONDARY OUTCOMES:
Overall response rate | 8 months
Complete response rate | 8 months
Progression-free survival | 3 years
Overall survival | 3 years
Quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Lukáš Smolej, M.D. Ph.D., Study Chair — Czech CLL Study Group
Locations (7):
- Czechia (7):
  - Department of Hematology - Oncology, University Hospital, Brno
  - Department of Hemato-Oncology, University Hospital, Olomouc
  - Department of Hematology, University Hospital, Pilsen
  - Department of Medicine - Hematology, University Hospital Kralovske Vinohrady, Prague
  - 1st Department of Medicine - Hematology, University General Hospital, Prague
  - Institute for Hematology and Blood Transfusion, Prague
  - 4th Department of Medicine - Hematology, University Hospital, Hradec Králové, ČR

REFERENCES:
- [Result] Smolej L. Therapy of elderly/comorbid patients with chronic lymphocytic leukemia. Curr Pharm Des. 2012;18(23):3399-405. doi: 10.2174/138161212801227096. PMID 22591390
- [Derived] Smolej L, Brychtova Y, Cmunt E, Doubek M, Spacek M, Belada D, Simkovic M, Stejskal L, Zygulova I, Urbanova R, Brejcha M, Zuchnicka J, Mocikova H, Kozak T; Czech CLL Study Group. Low-dose fludarabine and cyclophosphamide combined with rituximab in the first-line treatment of elderly/comorbid patients with chronic lymphocytic leukaemia/small lymphocytic lymphoma (CLL/SLL): long-term results of project Q-lite by the Czech CLL Study Group. Br J Haematol. 2021 May;193(4):769-778. doi: 10.1111/bjh.17373. Epub 2021 Feb 22. PMID 33618437
- See also: Czech CLL Study Group — http://www.cll.cz